CLINICAL TRIAL: NCT04774653
Title: Hypo-mineralization of Primary and Permanent Teeth in a Group of Children With Stunted Growth. A Cross Sectional Study.
Brief Title: Hypo-mineralization of Primary and Permanent Teeth in a Group of Children With Stunted Growth.A Cross Sectional Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Associate Professor Dr. Rania Abdallah Nasr, Associate Professor Dr. Rania Nasr, Cairo University
Other Study IDs: 00022021
Record Dates: First submitted 2021-02-19; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Short Stature; Hypomineralization Molar Incisor; Hypomineralization of Enamel
Keywords: MIH; HSPM; Stunded children; Prevalence
MeSH Terms: conditions — Dwarfism; Molar Hypomineralization; Dental Enamel Hypomineralization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MIH Group in short stature from 6-8 years old: Molar Incisor Hypomineralization in stunted children aged from 6-8 years
  Interventions: Other: No intervention
- HSPM Group in short stature from 5-8 years old: Hypomineralization of Second Primary Molars in stunted children aged from 5-8 years
  Interventions: Other: No intervention
- Both MIH &HSPM Group in stunted (from 5-8) years old: When both primary molars and permanent teeth( First permanent molars & permanent incisors) are hypo-mineralized in children with short stature with age range from 5-8 years old
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Associations and prevalence will be calculated

SUMMARY:
The second primary molar (SPM) development start at the same time as development of the first permanent molars (FPM) and permanent incisors so any systemic disturbance - causing stunted growth -occur , will result in hypo-mineralization of SPM as well as FPM and permanent incisors (Butler 1967, Weerheijm and Mejàre 2003).

The literature shows no previous studies that discuss the association between hypo- mineralized second primary molar (HSPM), MIH and the stunted growth in children.

aim: Estimate Prevalence of HSPM and MIH in stunted children.Evaluate the association between HSPM, MIH and the stunted growth in a group of Egyptian children.

• The diagnostic criteria for MIH established based on the European Academy of Pediatric Dentistry criteria (Weerheijm and Mejàre 2003) while diagnostic criteria for HSPM was established by (Elfrink et al. 2008).

DETAILED DESCRIPTION:
The second primary molar (SPM) development start at the same time as development of the first permanent molars (FPM) and permanent incisors so any systemic disturbance - causing stunted growth -occur , will result in hypo-mineralization of SPM as well as FPM and permanent incisors (Butler 1967, Weerheijm and Mejàre 2003).

The literature shows no previous studies that discuss the association between hypo- mineralized second primary molar (HSPM), MIH and the stunted growth in children.

aim: Estimate Prevalence of HSPM and MIH in stunted children.Evaluate the association between HSPM, MIH and the stunted growth in a group of Egyptian children.

. Methods of selection:

* Stunted children aged from 5 to 8 years attending outpatient clinic in Pediatric Dentistry Department, Faculty of Dentistry, Cairo University will be included in this study according to eligibility criteria.
* Informed consent will be obtained from children parents or guardians accepting to participate in the study. Medical and sociodemographic data will be recorded in patient chart.
* Children will be examined clinically on dental units using artificial light. Wet cotton swabs will be used to prior to examination to remove excess plaque or saliva.
* The diagnostic criteria for MIH established based on the European Academy of Pediatric Dentistry criteria (Weerheijm and Mejàre 2003) while diagnostic criteria for HSPM was established by (Elfrink et al. 2008).

Data sources and management:

Data will be obtained through clinical examination on participant children for MIH and HSPM according to the diagnosis criteria that we selected and the result will be collected in form of percentage for both conditions and the data will be analysis to show the relation between those conditions.

Handling of numerical/ quantitative variables:

Numerical data will be explored for normality by checking the data distribution, calculating the mean and median values and using Kolmogorov-Smirnov and Shapiro- Wilk tests. If the data was found to be normally distributed, it will be presented as mean and standard deviation values. If the assumption of normality was found to be violated, the data will be presented as median and range values.

Handling of categorical/ qualitative variables:

Categorical data will be represented as frequency (n) and percentage (%).

Statistical analysis:

Categorical data will be represented as frequency (n) and percentage (%) and will be analyzed using chi square test. Numerical data will be explored for normality by checking the data distribution, calculating the mean and median values and using Kolmogorov-Smirnov and Shapiro-Wilk tests. If the data was found to be normally distributed, it will be presented as mean and standard deviation values and independent t-test will be used for the analysis. The significance level will be set at P ≤0.05 for all tests. Statistical analysis will be performed with IBM® SPSS® Statistics Version 26 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* • Children aged from 5 to 8 years.

  * Both genders.
  * Stunted growth (Stunting: when the height for age is less than the mean by two standard deviations of the WHO Child Standards for growth or less than the 5th centile for age)

Exclusion Criteria:

* • Children with extracted primary second molars and permanent incisors and molars.

  * Children with history of dental trauma.
  * Children with orthodontic bands or dental appliances.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Egyptian children aged from 5 to 8 years with short stature attending to Outpatient Clinic of Pediatric Dentistry Department, Faculty of Dentistry, Cairo University.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HSPM in stunted children | 6 Months from April to October 2021
  Clinical examination (Weerheijm & Mejàre, 2003)
  Length /Height for age WHO growth charts (WHO, Length/Height for age Boys and Girls Available., www.who.int/childgrowth (2017).

SECONDARY OUTCOMES:
Prevalence of MIH in stunted children | 6 Months ( from April to October 2021)
  Clinical examination (Weerheijm & Mejàre, 2003) Length /Height for age WHO growth charts (WHO, Length/Height for age Boys and Girls Available., www.who.int/childgrowth (2017).

OTHER OUTCOMES:
Association of MIH &HSPM with short stature | 6 Months ( from April to October 2021)
  Is there an Association between HSPM, MIH and stunted growth in a group of Egyptian children?

CONTACTS AND LOCATIONS:
Overall Officials: Rania Nasr, Assoc. Prof., Principal Investigator — Department of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University
Locations (1):
- Department of Pediatric Dentistry, Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Informed consent Patient Diagnostic Chart Statistical Analysis